CLINICAL TRIAL: NCT01182103
Title: Epigenetic Regulation of Brain-Derived Neurotropic Factor (BDNF) in Patients With Major Depression
Brief Title: Epigenetic Regulation of BDNF in Major Depression
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tiao-Lai Huang, Head of Department of Psychiatry, Chang Gung Memorial Hospital
Other Study IDs: NSC99-2628-B-182-002-MY2
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Major Depressive Disorder
Keywords: Major depression; BDNF; DNA methylation; Histone modification
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major depressive patients
- Healthy subjects

SUMMARY:
The investigators will (1) detect the associations between brain-derived neurotrophic factor (BDNF) DNA methylation, histone modification, depressive symptoms, suicidal behavior and antidepressant responses in major depressive disorder (MDD) patients, (2) check the correlation between blood BDNF protein and RNA and BDNF rs6265 gene, and (3) discuss the possible mechanisms of epigenetic regulation of BDNF in Taiwanese major depressive patients.

DETAILED DESCRIPTION:
Brain-derived neurotrophic factor (BDNF) had been chosen as a candidate gene for a development of major depressive disorder (MDD). BDNF had been reported to have an important role on neuronal plasticity, axonal growth and connectivity, and participating in the local response to various types of neuronal stressors. BDNF also influences the differentiation of neurons.

In the past studies, the investigators had found that major depressive women had lower serum BDNF protein levels than healthy controls, and their BDNF levels became significantly increased after antidepressant treatments. In addition, some authors had found that reduced expression of BDNF was noted in postmortem brain of completed suicide subjects. Suicidal major depressive patients also had lower plasma BDNF levels than non-suicidal major depressive patients. These findings suggested that BDNF might play an important role in the suicidal behavior.

However, in past studies, the results did not fully explain why major depressive patients with same genotypes had different clinical expression, including the severity of depression, with/without suicide, and the treatment response. Recently, some papers found that there were relationships between epigenetic regulation, including DNA methylation and histone modification, and psychopathology of major depression. Therefore, we try to investigate the relationships between epigenetic regulation of BDNF and major depression.

ELIGIBILITY:
Inclusion Criteria:

The clinical screening and assessment in patients with major depression：

1. 40 major depression will be recruited in psychiatric inpatients according to DSM-IV criteria by a semi-structured interview. The assessment will be done by two senior psychiatrists. The intra-rater and inter-rater reliability will be done before this project started.
2. The patients had the ability to complete the written inform consent.
3. The choice of antidepressant drugs depended on the need of patients in natural treatment procedure. They included selective serotonin reuptake inhibitors (SSRI), eg. fluoxetine or paroxetine.
4. The 17-item Hamilton Depression Rating Scale (HAM-D) was used to assess severity of depression. The minimum baseline score of the 17-item HAM-D was 18.

Exclusion Criteria:

1. The patients had systemic diseases, including metabolic, heart, and liver diseases。
2. The patients had received any drugs before entering this protocol.
3. The patients were heavy smokers or dependent on alcohol.
4. The use of secondary generation anti-psychotic drugs and mood stabilizers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This 2-year study will be conducted in our clinical setting. By a semi-structured interview for DSM-IV criteria, a total of 160 subjectes (80 healthy controls and 80 patients with major depression) will be recruited in this study. In the first year (recruiting 40 healthy controls and 40 patients with major depression), the data of BDNF DNA methylation in all subjects will be collected. In the second year (recruiting another 40 healthy controls and 40 patients with major depression), the data of BDNF histone modification in all subjects will be collected and the mechanism of epigenetic regulation of BDNF in major depression will be discussed.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiao-Lai Huang, M.D., Principal Investigator — Chang-Gung Memorial Hospital, Kaohsiung
Locations (1):
- Department of Psychiatry, Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 1st, 2000 to July 31st, 2012, major depressive disorder patients were recruited from Kaohsiung Chang Gung Memorial Hospital, a tertiary medical center.
Period: Overall Study
Arm/Group | Major Depressive Patients | Healthy Subjects
Started | 48 | 62
Completed | 48 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Major Depressive Patients | Healthy Subjects | Total
Number analyzed (Participants) | 48 | 62 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 62 | 110
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.44 (12.09) | 30.18 (5.6) | 35.53 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 70
  Male | 16 | 24 | 40
Region of Enrollment [Number; unit: participants]
  Taiwan | 48 | 62 | 110

OUTCOME MEASURES:

1. Primary Outcome: Brain-derived Neurotrophic Factor (BDNF) DNA Methylation of Major Depressive Disorder (MDD) Patients and Healthy Controls
Description: averaged percentage of methylation at each CpG site listed
Time Frame: 2 years
Population: Only 39 out of the 48 MDD patients provided enough blood sample for this analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Major Depressive Patients | Healthy Subjects
Number analyzed (Participants) | 39 | 62
percent
  CpG site 24 | 92 (5.0) | 92 (3.0)
  CpG site 57 | 75 (5.4) | 75 (4.8)
  CpG site 80 | 65 (7.6) | 63 (6.2)
  CpG site 134 | 87 (4.2) | 86 (3.8)
  CpG site 140 | 49 (23.2) | 41 (24.7)
  CpG site 177 | 93 (3.9) | 94 (2.3)
  CpG site 203 | 88 (5.2) | 90 (2.9)
  CpG site 217 | 61 (8.0) | 51 (11.4)
  CpG site 324 | 95 (4.8) | 95 (2.4)
  CpG site 327 | 88 (4.7) | 90 (2.5)
  CpG site 345 | 97 (5.0) | 98 (3.0)
  CpG site 348 | 90 (6.0) | 91 (4.1)
  CpG site 362 | 89 (4.4) | 91 (2.0)
  CpG site 391 | 84 (4.8) | 85 (3.1)
Statistical Analysis 1: Comparison: Major Depressive Patients vs Healthy Subjects; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Histone Modification of MDD Patients Before and After Treatment and With Healthy Controls
Description: Chromatin immunoprecipitation (ChIP) was used to measure histone modification. The unit of our given machine is relative quantification, and a higher value indicated increased histone modification. The detailed method could be found in:
  Huebert DJ, Kamal M, O'Donovan A, Bernstein BE: Genome-wide analysis of histone modifications by ChIP-on-chip. Methods 2006; 40: 365-369.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: relative quantification
Arm/Group | Healthy Subjects | Major Depressive Patients Before Treatment | Major Depressive Patients After Treatment
Number analyzed (Participants) | 39 | 37 | 37
relative quantification
  BDNF promotor I acetyl-H3 | 3.5610 (2.79865) | .3124 (.53231) | .4321 (.32039)
  BDNF promotor I acetyl-H4 | 2.6346 (2.66175) | .3784 (.54543) | .4659 (.62056)
  BDNF promotor IV acetyl-H3 | 1.6356 (2.33692) | .4059 (.43157) | .4303 (.70365)
  BDNF promotor IV acetyl-H4 | 2.2795 (2.66175) | .4676 (.54543) | .4988 (.62056)
  BDNF promotor X acetyl-H3 | 3.8960 (1.94450) | .2564 (.36703) | .3640 (.34533)
  BDNF promotor X acetyl-H4 | 1.7433 (2.66175) | .2105 (.30502) | .2540 (.53050)
Statistical Analysis 1: Comparison: Healthy Subjects vs Major Depressive Patients Before Treatment vs Major Depressive Patients After Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Secondary Outcome: BDNF Levels of MDD Patients Before and After Treatment and Healthy Controls
Description: Serum BDNF levels were measured. MDD patients received antidepressant treatment, a standard biological management. Nothing novel (such as experimental drugs or management) is introduced in the treatment, so the research design is observational (of standard treatment).
  The choice of antidepressant drugs depended on the need of patients in natural treatment procedure. They included selective serotonin reuptake inhibitors (SSRI), eg. fluoxetine or paroxetine.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Healthy Subjects | Major Depressive Patients Before Treatment | Major Depressive Patients After Treatment
Number analyzed (Participants) | 62 | 48 | 48
ng/ml | 7.9386 (3.24400) | 5.6014 (4.46981) | 6.2803 (5.58535)
Statistical Analysis 1: Comparison: Healthy Subjects vs Major Depressive Patients Before Treatment vs Major Depressive Patients After Treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Major Depressive Patients | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/62
Other Adverse Events (participants affected / at risk) | 0/48 | 0/62

LIMITATIONS AND CAVEATS:
Limited funding prevented all samples from receiving all analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No